CLINICAL TRIAL: NCT03042442
Title: Relation Between Cachexia, Diabetes and periNeural Invasion in PANcreatic Cancer- Biomarkers Substudy
Acronym: CDNPAN
Status: Completed | Type: Observational
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Livia Petrusel, MD, PhD Student, Iuliu Hatieganu University of Medicine and Pharmacy
Other Study IDs: PCD 769/36
Record Dates: First submitted 2017-01-24; First posted 2017-02-03 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Pancreatic Cancer, Adult; Cachexia; Pain; Diabetes Mellitus
Keywords: pancreatic cancer; cachexia; perineural invasion; pain; diabetes
MeSH Terms: conditions — Pancreatic cancer, adult; Cachexia; Pain; Diabetes Mellitus; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples and pancreatic cancer tissue (from EUS FNA and surgery) will be collected from patients with pancreatic cancer adenocarcinoma at the time of diagnosis. The blood sample will be immediately prepared by centrifugation at 5000 × g for 5 min. The plasma samples were stored at -80 °C until use. Tissue will be embedded in paraffin.
  Point-of-care bio-markers will be assessed by using western blot analyses and immunohistochemistry.
  The participant will be explicitly asked for consent for storing the plasma sample.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with pancreatic cancer: Patients with pancreatic ductal adenocarcinoma, based on the results of an endoscopic ultrasonography (EUS) biopsy or surgery were enrolled at the diagnosis, before any therapeutic intervention.
  Interventions: Diagnostic Test: Point-of care biomarkers; Other: Clinical, venous blood samples, pancreatic tissue; Other: Follow-up
- health patients (controls): Health patients
  Interventions: Diagnostic Test: Point-of care biomarkers; Other: Clinical, venous blood samples, pancreatic tissue; Other: Follow-up

INTERVENTIONS:
Diagnostic Test: Point-of care biomarkers — Point-of care biomarkers(Activin,Midkine) assessed by WB and IHC
Other: Clinical, venous blood samples, pancreatic tissue — Clinical evaluation, venous blood samples and pancreatic tissue needed for determining point-of-care biomarkers.
Other: Follow-up — Participants will be assessed (by telephone) over a period of 2 years

SUMMARY:
The purpose of this study is to determine the interrelationship between cachexia, neural invasion and diabetes in patients with pancreatic cancer. Thus the investigators propose to identify the protein expression levels of Activin and Midkine in plasma of patients with different stages of pancreatic adenocarcinoma compared with healthy patients and to evaluate the possible correlation with diabetes, tumor size and tumor stage.

DETAILED DESCRIPTION:
In this study, the investigators will prospectively evaluate pancreatic adenocarcinoma patients with or without cachexia, perineural invasion and diabetes.

Patients with pancreatic ductal adenocarcinoma, based on the results of an endoscopic ultrasonography (EUS) biopsy or surgery were enrolled at the diagnosis and blood samples are drawn.

Thus the investigators propose to identify the protein expression levels of Activin and Midkine in plasma of patients with different stages of pancreatic adenocarcinoma compared with benign pancreatic disorders and healthy patients and to evaluate the possible correlation with diabetes, tumor size and tumor stage.

Furthermore, the investigators propose to identify the prognostic role of these biomarkers in the development of metastasis and survival in patients with adenocarcinoma, with and without diabetes and cachexia; to identify a new biomarker predictive of cachexia and eventually to select patients likely to benefit from treatment with antagonists of activin (or hypoglycemic treatment) and investigating the role of invasion neural in the appearance of cachexia in patients with pancreatic adenocarcinoma.

Follow-up: with phone-calls on an every 6 month, for up to 2 years, retaining the following data: survival, date of decease and its direct cause, the presence of tumor recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old
2. EUS or surgery biopsy confirming the diagnosis of adenocarcinoma
3. Informed consent

Exclusion Criteria:

1. obvious malabsorption
2. artificial nutrition
3. hyperthyroidism
4. major depression
5. other causes of malnutrition
6. refusing to enter the study

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatic ductal adenocarcinoma, based on the results of an endoscopic ultrasonography (EUS) biopsy or surgery were enrolled at the diagnosis, before any therapeutic intervention.
  Subjects of the study group were at least 18 years old, with no previous history of any other cancer in the last 5 years. Written consent was given prior to entry into the study.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of patients with loss of > 5% body weight | up to 6 months
  Using the BMI at admission and BMI at 6 months after admission

SECONDARY OUTCOMES:
Number of participants with pain as main symptom and antialgic therapy | up to 12 Months
  At baseline, throughout and at the end of the study as assessed by Visual Analogue Scale and type of antialgic treatment
Evaluation of Quality of Life of participants (EORTC QLQ-C30 ) | Change from baseline at 12 months
  At baseline, throughout and at the end of the study using EORTC QLQ-C30 questionnaire
Food intake assessment of participants using SNAQ questionnaire | Change from baseline at 6 months
  At baseline, throughout and at the end of the study using SNAQ questionnaire
Assessing the survival rate by phone-calls follow-up every 6 months, up to 2 years | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Livia Petrusel, MD, PhD, Principal Investigator — Iuliu Hatieganu University of Medicine
Locations (1):
- Regional Institute of Gastroenterology and Hepatology, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No